CLINICAL TRIAL: NCT05992506
Title: Electroencephalographic Biomarker to Predict the Development of Postoperative Delirium: a Protocol of an Observational Study in a Cohort of Patients From Five Centers
Brief Title: Electroencephalographic Biomarker to Predict Postoperative Delirium
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Instituto Nacional del Cancer, Chile (Unknown); Pontificia Universidad Catolica de Chile (Other); Hospital Base San Jose Osorno (Unknown); Clinica Santa Maria (Other)
Responsible Party: Sponsor
Other Study IDs: IT21I0041
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Delirium
Keywords: EEG; Postoperative Delirium; Risk Assessment; Anesthesia
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at risk of developing POD: * Patients older than 60 years
  * Scheduled for elective surgery of moderate or high risk (defined as that which requires a subsequent hospitalization of at least 3 days) under general anesthesia.
  * Signed informed consent.
  Interventions: Diagnostic Test: POD risk estimation using PEUMA

INTERVENTIONS:
Diagnostic Test: POD risk estimation using PEUMA — A software will analyze intraoperative EEG recording for the estimation of a POD Risk Index

SUMMARY:
Acute post-operatory cognitive dysfunction states are one of the most important complications in older patients that underwent surgery. Among them postoperative delirium (POD) is the the most studied. Patients who develop delirium have poorer long-term outcomes, such as longer length of hospital stay, institutionalization at discharge, and even higher mortality, and consequently, the human and economic costs significantly increase for the health system. Here the research team will use an observational cohort, investigator blinded in five-center with a primary endpoint to validate intraoperative EEG analysis as a reliable biomarker of postoperative delirium.

DETAILED DESCRIPTION:
Acute post-operatory cognitive dysfunction states are one of the most frequent complications in older patients after surgery, being POD the most important. Previous studies have shown than the incidence of POD in older patients range between 10-50%. Patients who develop POD have poorer long-term outcomes, such as longer length of hospital stay, institutionalization at discharge, and even higher mortality. Consequently, the human and economic costs associated to POD represents an important issue for health systems worldwide.

A key element to diminish POD and its burden on healthcare is early diagnostic. Current risk assessment tools are centered on clinical approaches based on cognitive tests (i.e., MoCA) and/or prediction models that uses patients' clinical variables (i.e., DELPHI score). We have developed a strategy that uses intraoperative EEG features as building blocks for a new POD risk assessment predictive model. This system, called PEUMA, uses data obtained from 95 patients from a previous study (NCT04214496).

This will be a multicenter (five-centers), observational study and its primary outcome will be PEUMA's ability to predict POD.

To calculate the sample size, the methodology described by Riley et al was used. This method is specially designed for clinical prediction models. Such a tool is available online (https://mvansmeden.shinyapps.io/BeyondEPV/). The parameters used were the following:

* Number of predictor candidates: 4
* Fraction of events: 0.22. 22% was used because it is the incidence of POD in the analysis of the preliminary data of the first stage and these are in the reporting range common worldwide.
* Estimation error of the classifier: 0.06. The authors suggest prediction errors small when evaluating binary outcomes (Yes POD/No POD) The calculation indicates a sample size of 240 patients. Considering a loss of 10% (in the preliminary results of the first stage the loss was 8%), the sample size is 264 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* Scheduled for high-risk elective surgery
* Need for at least 3 days of hospital stay after surgery
* Surgery performed under general anesthesia
* Written informed consent for participation in the trial

Exclusion Criteria:

* Patients with preoperative delirium or dementia
* Patients using neuroleptics drug during the past 6 months
* Patients with a history of encephalopathy, psychosis, stroke or brain trauma with neurologic sequels
* The use of ketamine or dexmedetomidine during surgery
* Emergency surgery
* Mechanical ventilation during the 72 after surgery
* Analphabetism
* Patients who do not talk Spanish
* Patients included in another clinical trial

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at risk of developing POD will be evaluated in the pre and postoperative period for cognitive dysfunction and the appearance of POD. In the intraoperative period, an EEG-based monitorization will be performed using a SedLine (Masimo, CA) Monitor.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Delirium | First 3 days after surgery
  Incidence of POD in the cohort diagnosed using the Confusion Assessment Method (CAM) twice/day

SECONDARY OUTCOMES:
Death | 30 days after surgery
  Number of deceased patients
Delirium Severity | First 3 days after surgery
  Delirium severity assessed by Cognitive Assessment Method - Severity (CAM-S)
Delirium Duration | First 3 days after surgery
  Duration of delirium during the postoperative period
Need for Mechanical Ventilation | First 3 days after surgery
  Number of patients that needed mechanical ventilation
Reintervention | First 3 days after surgery
  Number of patients who required other unanticipated surgery after the primary intervention
Unanticipated ICU hospitalization | First 3 days after surgery
  Number of patients that needed unanticipated intensive care unit (ICU) care

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan
  - Instituto Nacional del Cancer, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data might be shared with other researchers only if participants give written consent for that.

REFERENCES:
- [Result] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Result] Gutierrez R, Egana JI, Saez I, Reyes F, Briceno C, Venegas M, Lavado I, Penna A. Intraoperative Low Alpha Power in the Electroencephalogram Is Associated With Postoperative Subsyndromal Delirium. Front Syst Neurosci. 2019 Oct 18;13:56. doi: 10.3389/fnsys.2019.00056. eCollection 2019. PMID 31680886
- [Result] Wong CK, van Munster BC, Hatseras A, Huis In 't Veld E, van Leeuwen BL, de Rooij SE, Pleijhuis RG. Head-to-head comparison of 14 prediction models for postoperative delirium in elderly non-ICU patients: an external validation study. BMJ Open. 2022 Apr 8;12(4):e054023. doi: 10.1136/bmjopen-2021-054023. PMID 35396283